CLINICAL TRIAL: NCT01546727
Title: Clinic and Home Family Based Behavioral Treatment for Obese Preschoolers
Brief Title: Behavioral Treatment for Obese Preschoolers
Acronym: LAUNCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01DK091251 (NIH); 1R01DK091251-01A1 (NIH)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: Preschoolers; Obesity; Behavioral Treatment
MeSH Terms: conditions — Obesity | interventions — Spacecraft; Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Family Behavioral Treatment (Experimental): This intervention will provide nutritional counseling for a health diet, parent training in effective child behavioral management strategies, and stimulus control of the home environment delivered via group based clinic visits and individual home visits on alternate weeks
  Interventions: Behavioral: Behavioral Family Intervention
- Motivational Interviewing (Active Comparator): This intervention will shared information with parents about their child's weight and use motivational interviewing to elicit changes parents would like to make to their child diet and activity patterns.
  Interventions: Behavioral: Motivational Interviewing
- Standard of Care (No Intervention): Participants in this arm will be followed over time and be assessed on the primary and secondary outcomes at the same time points as the two treatment arms

INTERVENTIONS:
Behavioral: Behavioral Family Intervention — Three months of weekly treatment delivered via alternating group based clinic visits and individual home visits followed by three months of every other week treatment alternating between clinic and home.
  Other Names: LAUNCH
  Arms: Family Behavioral Treatment
Behavioral: Motivational Interviewing — Motivational interviewing will be delivered at the same frequency at the behavioral intervention with 4 in-person visits spaced at the first visit, month 3 and month 5. Phone calls will be conducted weekly during the first 3 months and every other week during months 4 through 6.
  Other Names: MI
  Arms: Motivational Interviewing

SUMMARY:
This study is a 3 arm, randomized, parallel group randomized clinical trial to test a clinic and home family behavioral intervention (LAUNCH) against 1) motivational interviewing (attention control; MI) and 2) standard of care (true standard of care control; STC) with 168 children ages 2 to 5 years who meet the criteria for obesity (>95th percentile for body mass index; BMI). Participants will be randomized to receive a 6 month intervention (LAUNCH, MI) or standard of care. The primary end-point will be change in BMI z-score at the end of treatment. The investigators will also assess maintenance of treatment gains at 6 and 12 months after treatment, and changes in factors thought to be mechanisms for change in weight (food intake and activity level), changes in the obesiogenic environment (parent weight, food intake and activity, and changes in the home food environment) and factors that could be negatively impacted (parent and child eating and feeding interactions).

DETAILED DESCRIPTION:
Obesity now affects an estimated 2.8 million children between the ages of 2 and 5 years, as the prevalence of obesity among preschool school age children has almost tripled from 5% of the population in 1971-1980 to 13.9% by 2004. Being obese at age 5 confers a 47 times greater risk of being overweight or obese at age 12. In fact being obese any time between 2 and 5 year increases the risk of remaining overweight or obese as an adult by four times the risk of nonobese preschoolers. Being obese as a preschooler also increases the risk of a number of serious health conditions, including a 2.6 times greater risk of developing type 2 diabetes by age 21 years. In fact, the obesity rate among preschoolers is thought to impose such a cumulative health risk across the life span that children born today, for the first time in history, are expected to have a shorter life expectancy than their parents by to 2 to 5 years. Early effective treatments for establish obesity during the preschool years have the potential to change the trajectory of obesity and related co-morbid health condition across the life-span by reducing obesity and changing the development of lifestyle habits of diet and exercise at a time when these are being formed. Yet research on interventions to reduce obesity in preschool children is severely limited and none exist that addresses established obesity in this age group. Therefore the current study has the potential to have a significant impact on public health by providing evidence-based treatment for obesity in preschoolers, a developmental period in which eating and activity patterns are being formed, that could significantly impact the trajectory of obesity thereby decreasing the population obesity rates and associated healthcare costs at across the life span. Fortunately, investigators are on their way to addressing the problem of obesity reduction in already obese preschoolers. The investigators have developed and conducted a pilot randomized clinical trial of a treatment program aimed at reducing obesity in already obese preschool children. The program (Learning about Activity and Understanding Nutrition for Child Health: LAUNCH) is tailored to the developmental stage of preschool children and produced promising preliminary results. In the proposed trial a 3 arm, randomized, parallel group design will test LAUNCH against 1) motivational interviewing (attention control; MI) and 2) standard of care (true standard of care control; STC) with 168 children ages 2 to 5 years who meet the criteria for obesity (>95th percentile for body mass index; BMI). Participants will be randomized to receive a 6 month intervention (LAUNCH, MI) or standard of care. The primary end-point will be change in BMI z-score at the end of treatment. The investigators will also assess maintenance of treatment gains at 6 and 12 months after treatment, and changes in factors thought to be mechanisms for change in weight (food intake and activity level), changes in the obesiogenic environment (parent weight, food intake and activity, and changes in the home food environment) and factors that could be negatively impacted (parent and child eating and feeding interactions).

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2 years 0 months to 5 years 11 months
* BMI percentile at or above the 95th percentile for age- and gender, but no more than 100% above the median BMI for age and gender.
* English-speaking
* Live within 50 miles of Cincinnati Children's Hospital Medical Center (CCHMC)
* Medical clearance from the child's pediatrician to participate.

Exclusion Criteria:

* Medical conditions known to promote obesity (e.g., Prader-Willi syndrome, Cushing's syndrome)
* Already involved with another weight control program
* Taking weight-affecting medications (e.g., steroids).
* A disability or illness that would preclude them from engaging in at least moderate intensity physical activity
* Developmental disability

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in BMIz score | Baseline to 6 months
  Body Mass Index z-score

SECONDARY OUTCOMES:
Change in BMI z at follow up | Baseline, 6 months, 12 months, 18 months
Change in Caloric Intake | Baseline, 6 months, 12 months, 18 months
  Three 24 hour dietary recalls at each time point
Change in Physical Activity | Baseline, 6 months, 12 months, 18 months
  Physical Activity will be measured using Accelermeters set in 15 sec epochs
Change in home health environment | Baseline, 6 months, 12 months, 18 months
  Home observation recording of food (e.g.,fruits, vegetables, high calorie foods and beverages)and presence of TV in child's bedroom
Changes in parent calorie intake | Baseline, 6 months, 12 months, 18 months
  Will assess using Block 2005 Food Frequency
Changes in parent physical activity | Baseline, 6 months, 12 months, 18 months
  Will be assessed using the Paffenbarger Activity Questionnaire for calorie expenditure
Parenting and Child Eating Behaviors | Baseline, 6 month, 12 months, 18 months
  Will assess using Parenting Styles and Dimensions, About Your Child's Eating - Revised, and Child Feeding Questionnaire
Change in Health Related Quality of Life | Baseline, 6 months, 12 months, 18 months
  Will be assessed using the PedQL

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Stark, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Stark LJ, Filigno SS, Kichler JC, Bolling C, Ratcliff MB, Robson SM, Simon SL, McCullough MB, Clifford LM, Stough CO, Zion C, Mara CA. Maintenance Following a Randomized Trial of a Clinic and Home-based Behavioral Intervention of Obesity in Preschoolers. J Pediatr. 2019 Oct;213:128-136.e3. doi: 10.1016/j.jpeds.2019.05.004. Epub 2019 Jun 21. PMID 31230889
- [Derived] Robson SM, Ziegler ML, McCullough MB, Stough CO, Zion C, Simon SL, Ittenbach RF, Stark LJ. Changes in diet quality and home food environment in preschool children following weight management. Int J Behav Nutr Phys Act. 2019 Feb 4;16(1):16. doi: 10.1186/s12966-019-0777-6. PMID 30717746
- [Derived] Stark LJ, Spear Filigno S, Bolling C, Ratcliff MB, Kichler JC, Robson SM, Simon SL, McCullough MB, Clifford LM, Odar Stough C, Zion C, Ittenbach RF. Clinic and Home-Based Behavioral Intervention for Obesity in Preschoolers: A Randomized Trial. J Pediatr. 2018 Jan;192:115-121.e1. doi: 10.1016/j.jpeds.2017.09.063. Epub 2017 Nov 14. PMID 29150147
- [Derived] Stark LJ, Filigno SS, Bolling C, Ratcliff MB, Kichler JC, Robson SL, Simon SL, McCullough MB, Clifford LM, Stough CO, Zion C, Ittenbach RF. Learning about Activity and Understanding Nutrition for Child Health (LAUNCH): Rationale, design, and implementation of a randomized clinical trial of a family-based pediatric weight management program for preschoolers. Contemp Clin Trials. 2017 Jan;52:10-19. doi: 10.1016/j.cct.2016.10.007. Epub 2016 Oct 21. PMID 27777128
- [Derived] Robson SM, Bolling C, McCullough MB, Stough CO, Stark LJ. A Preschool Obesity Treatment Clinical Trial: Reasons Primary Care Providers Declined Referrals. J Pediatr. 2016 Oct;177:262-266.e1. doi: 10.1016/j.jpeds.2016.06.027. Epub 2016 Jul 22. PMID 27453375